CLINICAL TRIAL: NCT03763994
Title: Reliability of an Objective Measurement to Assess Lumbar Spine Motion in Healthy Controls and in Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. Christoph Maier, Pain Medicine, Ruhr University of Bochum
Other Study IDs: 4385-12
Record Dates: First submitted 2012-12-20; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Reliability, Validity of Measurement to Assess Lumbar Spine Motion; Comparison of Healthy Subjects and Low Back Pain Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control group 1: Never low back pain in the last 3 months
- Control group 2: occasionally (1-30days) low back pain in the last 3 months
- Low back pain group 3: frequently (31-60days) low back pain in the last 3 months
- Low back pain group 4: daily (61-90days) low back pain in the last 3 months

SUMMARY:
Main of the study is to assess the reliability of a new objective tool to measure lumbar spine motion. The data will be collected from healthy subjects and subjects with frequent or daily low back pain in the last three months. In addition we compare the results of the motion measurements with disability and pain questionnaires such as the Roland Morris, Oswestry Disability Index and the Brief Pain Inventory.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years, informed consent, sufficient German skills <30 days low back pain in the last 90 days (control group) >31days of low back pain in the last 90 days (low back pain group)

Exclusion Criteria:

* neurological disorder (including multiple sclerosis, Stroke, Parkinson´s disease), Current pain >= 4 (NSR)/intake of analgesic in the last 24h/ previous low back surgery (control group), inability to perform choreography (LBP group)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Low back pain patients were recruited among in-and outpatients of the Department of Pain Medicine at the Bergmannsheil, Bochum. The subjects of the control groups were recruited by distributing flyers in sport groups and among hospital staff and friends.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
reliability of measurement tool | February 2012-February 2013
  reliability of measurement tool

CONTACTS AND LOCATIONS:
Locations (1):
- Berufsgenossenschaftliches Universitätklinikum Bergmannsheil, Bochum, Northrine-Westfalia, Germany